CLINICAL TRIAL: NCT06289660
Title: Multicenter Italian Observational Cohort Study on Tuberculosis in Pediatric Age
Brief Title: Multicenter Italian Cohort Study on Tuberculosis in Pediatric Age
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Luisa Galli, Clinical Professor, Meyer Children's Hospital IRCCS
Other Study IDs: PED-TB22
Record Dates: First submitted 2024-02-15; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the WHO report of 2021, approximately 10 million new cases were reported in 2020, of which 1 million occurred in the pediatric population. However, epidemiological data available on tuberculosis (TB) in pediatric age are extremely limited due to diagnostic challenges in this patient category. Furthermore, children are almost never included in national surveillance systems due to the lack of connections between individual pediatricians, pediatric hospitals, and national surveillance programs. It is therefore reasonable to assume that the disease may be significantly underestimated both in Italy and worldwide.

DETAILED DESCRIPTION:
In recent decades, Tuberculosis (TB) has been considered, in industrialized countries, as predominantly an infectious disease of the elderly. However, since the 2000s, TB has re-emerged not only in the elderly but also in the young and especially in pediatric populations. Among the factors influencing the increase in the incidence of this pathology are certainly to be considered the rise in immigration from countries with high endemicity, where TB still represents a significant cause of morbidity and mortality, the spread of immunodeficiency caused by HIV infection, the use of immunosuppressive drugs, and the emergence of strains of M. tuberculosis resistant to traditional antibiotic therapy.

According to the WHO report of 2021, approximately 10 million new cases were reported in 2020, of which 1 million occurred in the pediatric population. However, epidemiological data available on TB in pediatric age are extremely limited due to diagnostic difficulties in this patient category. In children, in fact, bacteriological examination is negative in 95% of cases, and the diagnosis is made through a combination of clinical criteria and tests that are poorly specific for tuberculous infection and especially not universally accepted. In addition to diagnostic controversies, children are almost never included in national surveillance systems due to the lack of connections between individual pediatricians, pediatric hospitals, and national surveillance programs. It is therefore reasonable to assume that this condition may be significantly underestimated both in Italy and worldwide.

Another important aspect to consider is that tuberculous disease, whether active or latent, in a child should be considered a sentinel event that indicates recent transmission of M. tuberculosis within the community. Especially in the pediatric population, in addition to the mandatory reporting of confirmed cases of TB disease, it is important to identify cases of latent TB through historical and diagnostic criteria. Children indeed have a greater likelihood that the disease will progress to the active form compared to adults and that the progression will be towards a more severe form. Children with latent tuberculous infection also become a reservoir for the transmission of the infection, fueling future epidemics.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (0-18 years old) at the time of the initial observation
* Patients affected by active and latent TB, as defined by the criteria of the World Health Organization
* Patients exposed to TB who are found to be non-infected at the end of the window period
* Informed consent signed by parents/legal guardian or by the patient who has reached the legal age of consent, assent of the minor

Exclusion Criteria:

* None

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: During the study, data will be collected on patients affected by active TB, latent TB, and TB-exposed non-infected individuals from each participating center. The study will take place at the main pediatric centers in Italy that consecutively admit patients diagnosed with active and latent TB, as well as individuals exposed to tuberculosis who are seen at participating clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2033-01-02 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of Tuberculosis | Baseline-pretreatment, through treatment period completion, an average of 6 months, outcome at 24 months
  Describe the epidemiology of pediatric tuberculosis in the country also for the definition of control and prevention measures.

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - Meyer Children's Hospital IRCCS, Florence, Firenze
  - Ospedale Pediatrico Giovanni XXIII, Bari
  - Ospedale di Belluno, Belluno
  - Università di Bologna, Bologna
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore, Policlinico, Milan
  - Ospedale Luigi Sacco, Milan
  - Policlinico di Modena, Modena
  - Università Federico II, Napoli
  - Ospedale dei Bambini "G.Di Cristina", Palermo
  - Ospedale di Parma, Parma
  - IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda USL Toscana Centro, Prato
  - IRCCS Ospedale Pediatrico Bambin Gesù, Roma
  - Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Ospedale Regina Margherita, Torino

IPD SHARING:
Plan to Share IPD: No